CLINICAL TRIAL: NCT04515823
Title: The Flat OGTT During Pregnancy -Prevalence and Risk for Adverse Outcomes
Brief Title: Flat OGTT (Oral Glucose Tolerance Test) During Pregnancy
Status: Completed | Type: Observational
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0052-20-HYMC
Record Dates: First submitted 2020-08-13; First posted 2020-08-17 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Pregnancy Related

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to examine the relationship between "flat" sugar curve on OGTT-glucose tolerance test during pregnancy, neonatal birthweight and other perinatal outcomes.

DETAILED DESCRIPTION:
A retrospective cohort analysis of all women delivered in one university affiliated medical center between January 1st 2018 and December 31th 2019 with documented 100 grams OGTT results.

ELIGIBILITY:
Inclusion Criteria:

* Performing the OGTT test during the pregnancy

Exclusion Criteria:

* lack of documentation or Non-performance of OGTT test during the pregnancy.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All women delivered in one university affiliated medical center between January 1st 2018 and December 31th 2019 with documented 100 grams OGTT results.
Sampling Method: Probability Sample
Enrollment: 2085 (Actual)
Dates: Start 2020-04-26 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the characteristics and perinatal outcomes of parturients with a flat glucose curve on 100 grams oral glucose tolerance test (OGTT). | 10 months
  A flat OGTT curve occurs in a younger, leaner population. Although flat OGTT can possibly reflect some degree of hyperinsulinemia, it is generally not associated with adverse maternal or neonatal outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Rinat Gabbay-Benziv, M.D, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Department of Obstetrics and Gynecology, Hillel-Yaffe Medical Center, Hadera, Israel